CLINICAL TRIAL: NCT01933503
Title: An Open Label, Randomized, Single Dose and Multiple Dose Trial to Assess the Pharmacokinetics of Obeticholic Acid (OCA)
Brief Title: Single Dose and Multiple Dose Trial to Assess Pharmacokinetics of Obeticholic Acid (OCA)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Intercept Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 747-105
Record Dates: First submitted 2013-08-28; First posted 2013-09-02 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-12

CONDITIONS: Healthy
Keywords: MAD; SAD; Obeticholic Acid (OCA)
MeSH Terms: interventions — obeticholic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- OCA 5 mg (Experimental): OCA 5 mg, 1 mg by mouth followed by 2 days of no investigational product (IP); then OCA 5 mg by mouth for 14 days.
  Interventions: Drug: OCA 5 mg
- OCA 10 mg (Experimental): OCA 10 mg, 1 mg by mouth followed by 2 days of no investigational product (IP); then OCA 10 mg by mouth for 14 days.
  Interventions: Drug: OCA 10 mg
- OCA 25 mg (Experimental): OCA 25 mg, 1 mg by mouth followed by 2 days of no investigational product (IP); then OCA 25 mg by mouth for 14 days.
  Interventions: Drug: OCA 25 mg

INTERVENTIONS:
Drug: OCA 5 mg
  Other Names: INT-747; 6α-ethyl chenodeoxycholic acid; 6-ECDCA
  Arms: OCA 5 mg
Drug: OCA 10 mg
  Other Names: INT-747; 6α-ethyl chenodeoxycholic acid; 6-ECDCA
  Arms: OCA 10 mg
Drug: OCA 25 mg
  Other Names: INT-747; 6α-ethyl chenodeoxycholic acid; 6-ECDCA
  Arms: OCA 25 mg

SUMMARY:
This is a single center, open label, randomized, parallel design, single and multiple dose trial to evaluate the pharmacokinetics(PK), safety and tolerability of obeticholic acid (OCA).

DETAILED DESCRIPTION:
Twenty-four eligible subjects will be enrolled and randomized to 1 of 3 treatment groups (5 mg, 10 mg, or 25 mg) in a treatment ratio of 1:1:1 and no less than a ratio of 1:1 for female: male subjects. The study comprises single dose and multiple dose phases. The randomized dose administered in the single dose phase will be the subject's dose level for the multiple dose phase. A single dose of OCA (5 mg, 10 mg, or 25 mg) will be administered on Day 1. PK, safety, and tolerability will then be assessed for 3 days. On Day 4, the multiple dose phase will begin at the same dose level (5 mg, 10 mg, or 25 mg), with subjects receiving OCA once daily for 14 days. PK, safety, and tolerability will be assessed for 2 weeks at the clinical site following the last investigational product (IP) dose on Day 17. Subjects will be confined at the inpatient trial site from Day 0 until the morning of Day 30. They will return to the study site on Day 37 for follow up.

ELIGIBILITY:
Subjects are required to meet the following criteria in order to be included in the trial.

1. Males or females age 18 to 55 years
2. Contraception: Oral contraceptives are not allowed to be used for 2 weeks prior to trial start, during the trial, and for 30 days after the last dose of OCA. Therefore, female subjects must be postmenopausal, surgically sterile, or if premenopausal, be prepared to use more than 1 effective (≤ 1% failure rate) method of contraception during the trial and until at least 30 days after the last dose of OCA. Effective methods of contraception for males and females are considered to be the following:

   1. Double barrier method, ie, (i) condom, with spermicide (male or female) or (ii) diaphragm with spermicide
   2. Intrauterine device (IUD)
   3. Vasectomy (partner)
3. Good general health as determined by medical history and by results of physical exam, vital signs, ECG, and clinical laboratory tests obtained within 14 days prior to IP administration
4. Body mass index (BMI) between 18 and 30 kg/m2; BMI is determined by the following equation: BMI = weight/height2 (kg/m2).
5. Willing to abstain from alcohol, caffeine, and xanthine containing food and beverages for 72 hours prior check in and during participation of the inpatient period of the trial
6. Willing and able to give written informed consent

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from the trial:

1. Prior exposure to OCA (INT-747; 6-ECDCA)
2. History of known or suspected clinically significant hypersensitivity to OCA or any of its components
3. History or presence of any disease or condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs including bile salt metabolism in the large intestine, eg, inflammatory bowel disease (IBD)
4. History of gastrointestinal surgeries or gall bladder removal (cholecystectomy)
5. History or presence of a clinically significant cardiovascular, hepatic, diabetic, gastrointestinal, metabolic, neurologic, pulmonary, endocrine, psychiatric, or neoplastic disorder(s)
6. History of known or suspected clinically significant hypersensitivity to any drug, aside from penicillin
7. Ingestion of a prescription medication, including oral contraceptives and bile acid sequestrants, within 14 days prior to IP dosing or ingestion of an over the counter medication within 7 days prior to IP dosing
8. Participation in radiologic examinations involving parenteral administration of iodinated contrast materials within 2 weeks prior to screening, or subsequently through the end of trial participation
9. History or presence of alcohol abuse (defined as consumption of more than 210 mL of alcohol per week, or the equivalent of fourteen 4 ounces [oz] glasses of wine or fourteen 12 oz. cans/bottles of beer or wine coolers per week) or positive alcohol tests
10. History or presence of substance abuse within the past 2 years or positive drug screen tests
11. Smoker or use of any tobacco or nicotine containing products
12. Any screening laboratory test for which the results are not within the normal reference range and considered clinically significant
13. Participation in another investigational drug trial within 30 days prior to Day 0
14. History of noncompliance to medical regimens, or subjects who are considered to be potentially unreliable
15. Blood or plasma donation within 30 days prior to Day 0
16. Mental instability or incompetence
17. Presence of human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus (HBV) at screening
18. Known or suspected Pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax observed) | 3 days - single dose, 33 days - Multi dose
  Maximum concentration (observed) following single and multiple doses of OCA 5 mg, 10 mg, and 25 mg
Time to maximum concentration (tmax) | 3 days - single dose, 33 days - Multi dose
  Time to maximum concentration (tmax)
Area under the concentration vs. time curve (AUCt) | 3 days - single dose, 33 days - Multi dose
  Area under the concentration vs. time curve (AUCt) from time 0 to the last sampling time with measurable analyte concentration, calculated by the linear trapezoidal method
Area under the concentration vs. time curve from time 0 to 24 hours (AUC0-24) | 24 hours
  Area under the concentration vs. time curve from time 0 to 24 hours (AUC0-24) with measurable analyte concentration, calculated by the linear trapezoidal method
The ratio of each conjugate to OCA | 3 days - single dose, 33 days - Multi dose
  The ratio of each conjugate to OCA for exposure PK parameters for both single and multiple dose assessments.
Accumulation ratios (Rac) based on AUC, Cmax and Cmin | 17 days
  Accumulation ratios (Rac) based on AUC, Cmax and Cmin will be calculated for OCA and its conjugates (glyco-OCA and tauro-OCA) from Day 1 to Day 17

CONTACTS AND LOCATIONS:
Overall Officials: David Shaprio, M.D., Study Director — Intercept Pharmaceuticals, San Diego, CA 92122
Locations (1):
- Spaulding Clinical Research, West Bend, Wisconsin, United States

REFERENCES:
- [Derived] Friedman ES, Li Y, Shen TD, Jiang J, Chau L, Adorini L, Babakhani F, Edwards J, Shapiro D, Zhao C, Carr RM, Bittinger K, Li H, Wu GD. FXR-Dependent Modulation of the Human Small Intestinal Microbiome by the Bile Acid Derivative Obeticholic Acid. Gastroenterology. 2018 Dec;155(6):1741-1752.e5. doi: 10.1053/j.gastro.2018.08.022. Epub 2018 Aug 23. PMID 30144429
- [Derived] Edwards JE, LaCerte C, Peyret T, Gosselin NH, Marier JF, Hofmann AF, Shapiro D. Modeling and Experimental Studies of Obeticholic Acid Exposure and the Impact of Cirrhosis Stage. Clin Transl Sci. 2016 Dec;9(6):328-336. doi: 10.1111/cts.12421. Epub 2016 Oct 15. PMID 27743502